CLINICAL TRIAL: NCT05075434
Title: Effects of the Diacutaneous Fibrolysis Approach on Gastrocnemius Length, Plantar Fascia Viscoelasticity and Plantar Arch Diameters in Patients With Plantar Fasciitis.
Brief Title: Effects of the Diacutaneous Fibrolysis Approach in Patients With Plantar Fasciitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER-2021-A1
Record Dates: First submitted 2021-09-28; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Plantar Fascitis; Heel Pain Syndrome
Keywords: plantar fasciitis; diacutaneous fibrolysis; primary care; plantar arch
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive the protocol prescribed by the health centre (calf stretching exercises, plantar fascia, proprioception exercises, ultrasound, magnet therapy and gait re-education and proprioceptive exercises for 40-45 minutes). In addition, you will receive 15 minutes of the instrumental technique of diacutaneous fibrolysis. Participants will receive 8 treatment sessions spread over 4 weeks (2 sessions per week).
  Interventions: Other: Conventional Treatment; Other: Diacutaneous fibrolysis
- Control Group (Active Comparator): This protocol will be the one prescribed by the health centre. It consists of calf stretching exercises, plantar fascia, proprioceptive exercises, ultrasound, magnetic therapy and gait re-education and proprioceptive exercises for 40-45 minutes. Participants will receive 8 treatment sessions spread over 4 weeks (2 sessions per week).
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Conventional Treatment — This protocol will be the one prescribed by the health centre. It consists of calf stretching exercises, plantar fascia, proprioceptive exercises, ultrasound, magnetic therapy and gait re-education and proprioceptive exercises for 40-45 minutes. Participants will receive 8 treatment sessions spread over 4 weeks (2 sessions per week).
Other: Diacutaneous fibrolysis — 15 minutes of the treatment technique. The FD intervention will be carried out with the same duration and protocol for all participants.
  The intervention protocol will be: Start with the point of maximum tension between the two muscle bellies of the calf and hamstring (reverse hook). Then work on the peroneus longus lateralis and soleus. Then the external calf muscle belly and soleus and the internal calf muscle belly and soleus. Then work on the tendon of the flexor hallucis proprio of the big toe and the inner edge of the Achilles tendon and peroneus longus. Then treatment of the peroneus longus with the peroneus brevis. Scraping of the insertion of the Achilles tendon, hooking of the internal and external part of the plantar fascia. Finally, longitudinal friction of the plantar fascia.
  Arms: Intervention Group

SUMMARY:
Diacutaneous Fibrolysis (FD) is a physiotherapy technique based on Cyricax's transverse massage. Kurt Ekman, its creator, observed that Cyriax's deep transverse massage was intended to achieve a mechanical effect on the tissues, but this had a series of disadvantages such as the difficulty in penetrating between tissue septa due to the large surface area of the finger tips, as well as its soft consistency in the face of adhesions or fibrosis.

Hypothesis: Adding FD to the gastrocnemius and plantar fascia to a primary care treatment protocol will produce a decrease in the stiffness (viscoelastic property) of the plantar fascia, an increase in length, width, height and a decrease in the plantar arch, as well as an increase in the length of the gastrocnemius greater than not adding it in subjects with plantar fasciitis.

Data collection. Once the participant has passed the selection criteria and signed the informed consent form, the measurements of the anthropometric variables and classification of the foot with the Foot Posture Index will be carried out. Subsequently, the dependent variables will be collected, starting with active and passive gastrocnemius flexibility, followed by measurements with the anthropometric foot measurement platform (foot length, arch height in loading and unloading, arch height index, foot width in loading and unloading, windlass force at 20º, 40º and maximum, myotonometry measurements (tone, stiffness, elasticity, relaxation and creep) and pain. Once the initial variables have been recorded, the first patient intervention will be carried out according to the assigned group. A total of 8 sessions will be carried out over 4 weeks (2 sessions per week). The variables of this study will be collected at the beginning of the study and at the end of the 8 intervention sessions (1 month).

Intervention "Protocol The usual protocol that the health service guidelines for this pathology will be carried out. The protocol consists of calf stretching exercises, plantar fascia, proprioception exercises, ultrasound, magnet therapy and gait re-education and proprioceptive exercises. The average intervention lasts between 30-45 minutes.

"Protocol "+FD Participants in this group will additionally receive 15 minutes of the treatment technique.

The FD intervention will be carried out with the same duration and protocol for all participants.

The intervention protocol will be: Start with the point of maximum tension between the two muscle bellies of the calf and hamstring (Reverse hook). Then work on the peroneus longus lateralis and soleus. Then the external calf muscle belly and soleus and the internal calf muscle belly and soleus. Then work on the tendon of the flexor hallucis proprio of the big toe and the inner edge of the Achilles tendon and peroneus longus. Then treatment of the peroneus longus with the peroneus brevis. Scraping of the insertion of the Achilles tendon, hooking of the internal and external part of the plantar fascia. Finally, longitudinal friction of the plantar fascia.

The participant will be in prone position with a support on the front of the leg with the foot off the stretcher. The physiotherapist will be in a standing position next to the participant. The procedure will be to palpate the different intermuscular septa and grooves and then perform the FD phases with the hook (supplementary transverse traction).

DETAILED DESCRIPTION:
Diacutaneous Fibrolysis (FD) is a physiotherapy technique based on Cyricax's transverse massage. Kurt Ekman, its creator, observed that Cyriax's deep transverse massage was intended to achieve a mechanical effect on the tissues, but this had a series of disadvantages such as the difficulty in penetrating between tissue septa due to the large surface area of the finger tips, as well as its soft consistency in the face of adhesions or fibrosis.

To overcome these difficulties, Ekman designed hooks that allowed, according to Ekman himself, to treat areas located in depth. The hooks used in the current FD are metallic, curved at both ends, which allow working more specifically in depth and transversally to the tissue without slipping on the skin, focusing the mechanical effect and reducing the stress on the physiotherapist.

Its mechanical effect is described as the elimination of areas of fibrosis, trying to recover physiological sliding between tissue planes, and although there is little scientific evidence on the mechanical effects of FD, several authors have described clinical modifications in passive muscle resistance to stretching or gains in joint movement. These modifications suggest a tendon mechanical adaptation as suggested by Lévenez, Guissard and Duchateau. A cutaneous circulatory effect is also described and is the most visible effect achieved with instrumental soft tissue mobilisation techniques. In addition, Burnotte and Duby, observed that venous return was improved with FD in several pathologies, although the mechanism is unknown. Histamine released after FD application is thought to be responsible for these effects. Neurophysiological effects were observed by Veszely et al. in the application of FD to the triceps suralis, in which neuromodulatory effects were observed 30 minutes after application, with a decrease in tendon reflexes. A neuromuscular effect has now also been described in response to tensomiography and myotonometry with a decrease in tone and stiffness of the triceps suralis muscle in asymptomatic subjects, which was maintained 30 minutes post-intervention.

The relationship of the gastrocnemius with the plantar fascia and this with the maintenance of the plantar arch is well known. The gastrocnemius, with the continuation of the Achilles tendon, modulates the tension of the plantar aponeurosis. As the tension of the triceps suralis increases, so does the tension of the plantar fascia. This is very important for weight-bearing transition during gait. The direction of the tendons of the extrinsic muscles of the foot shows their ability to provide dynamic support and control of the longitudinal and transverse components of the plantar arch. The global movements will provide both absorption and propulsive capacity during dynamic activities.

Plantar fasciitis is one of the most common foot disorders, being the leading cause of heel pain in primary care and accounting for 80% of all heel pain. Plantar fasciitis is a common injury caused by repetitive traction of the origin of the plantar fascia on the distal calcaneus.

In clinical practice, the gastrocnemius approach is commonly used to treat plantar fascia and Achilles problems. FD is one of the techniques used for these treatments; however, no studies have been found on its clinical effects or the effects of this technique on the plantar arch.

Hypothesis: Adding FD to the gastrocnemius and plantar fascia to a primary care treatment protocol will produce a decrease in the stiffness (viscoelastic property) of the plantar fascia, an increase in length, width, height and a decrease in the plantar arch, as well as an increase in the length of the gastrocnemius greater than not adding it in subjects with plantar fasciitis.

Data collection. Once the participant has passed the selection criteria and signed the informed consent form, the measurements of the anthropometric variables and classification of the foot with the Foot Posture Index will be carried out. Subsequently, the dependent variables will be collected, starting with active and passive gastrocnemius flexibility, followed by measurements with the anthropometric foot measurement platform (foot length, arch height in loading and unloading, arch height index, foot width in loading and unloading, windlass force at 20º, 40º and maximum, myotonometry measurements (tone, stiffness, elasticity, relaxation and creep) and pain. Once the initial variables have been recorded, the first patient intervention will be carried out according to the assigned group. A total of 8 sessions will be carried out over 4 weeks (2 sessions per week). The variables of this study will be collected at the beginning of the study and at the end of the 8 intervention sessions (1 month).

Intervention "Protocol The usual protocol that the health service guidelines for this pathology will be carried out. The protocol consists of calf stretching exercises, plantar fascia, proprioception exercises, ultrasound, magnet therapy and gait re-education and proprioceptive exercises. The average intervention lasts between 30-45 minutes.

"Protocol "+FD Participants in this group will additionally receive 15 minutes of the treatment technique.

The FD intervention will be carried out with the same duration and protocol for all participants.

The intervention protocol will be: Start with the point of maximum tension between the two muscle bellies of the calf and hamstring (Reverse hook). Then work on the peroneus longus lateralis and soleus. Then the external calf muscle belly and soleus and the internal calf muscle belly and soleus. Then work on the tendon of the flexor hallucis proprio of the big toe and the inner edge of the Achilles tendon and peroneus longus. Then treatment of the peroneus longus with the peroneus brevis. Scraping of the insertion of the Achilles tendon, hooking of the internal and external part of the plantar fascia. Finally, longitudinal friction of the plantar fascia.

The participant will be in prone position with a support on the front of the leg with the foot off the stretcher. The physiotherapist will be in a standing position next to the participant. The procedure will be to palpate the different intermuscular septa and grooves and then perform the FD phases with the hook (supplementary transverse traction).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Medical diagnosis of plantar fasciitis.
* Sign the informed consent for participation in the study.

Exclusion Criteria:

* Present pathology in the lower limbs other than plantar fasciitis, which may alter the assessments.
* History of orthopaedic injuries in the last 6 months that may influence correct standing.
* Use of corrective insoles due to plantar arch problems.
* Skin lesions in the region of application that prevent the application of the technique.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Foot Posture Index (score) | Change between baseline(immediately before intervention) and post intervention (1 month)
  Is a clinical diagnostic tool that uses observation and palpation of clinical criteria to classify the posture of the loaded foot. It consists of 6 items, each of which is scored from -2 to +2, with 0 being the neutral value of the foot and the total score ranging from -12 to +12. The assessment is carried out with the patient standing upright in a relaxed position.
Anthropometric foot measurement platform (p-MAC) (milimeters) | Change between baseline(immediately before intervention) and post intervention (1 month)
  Is a platform for measuring three variables: total foot length, truncated length (length to the head of the first metatarsal) and the height of the dorsal arch.
Myotonometry (Hz) | Change between baseline(immediately before intervention) and post intervention (1 month)
  Myotonometry is a non-invasive tool that assesses the viscoelastic properties of muscle, fascia and connective tissue. Muscle tone (Hz): is defined as the intrinsic tension of the muscle at the cellular level in the resting state.
Myotonometry (N/m) | Change between baseline(immediately before intervention) and post intervention (1 month)
  Myotonometry is a non-invasive tool that assesses the viscoelastic properties of muscle, fascia and connective tissue. Stiffness (N/m): The biomechanical property of the muscle that characterises the resistance to an external force that deforms its initial shape.
Myotonometry (m/s) | Change between baseline(immediately before intervention) and post intervention (1 month)
  Myotonometry is a non-invasive tool that assesses the viscoelastic properties of muscle, fascia and connective tissue. Relaxation (m/s): The time it takes for a muscle to regain its shape after the removal of an external force.

SECONDARY OUTCOMES:
Active Gastrocnemius Flexibility (º) | Change between baseline(immediately before intervention) and post intervention (1 month)
  The range of motion of active ankle dorsiflexion shall be assessed with the Lunge test. The test shall be performed by placing the foot perpendicular to a wall and throwing the knee towards the wall. The foot is moved away from the wall until the maximum range of dorsiflexion is reached. To ensure that the heel does not lift off the ground, the examiner shall place a band under the heel and apply tension.
Pasive Gastrocnemius Flexibility (º) | Change between baseline(immediately before intervention) and post intervention (1 month)
  To assess passive gastrocnemius flexibility, volunteers will be placed in the supine shirt with the foot relaxed. An inclinometer shall be placed on the plantar surface of the foot in the initial relaxed position of ankle dorsiflexion, placing the inclinometer in the 0-value position. A progressive force shall be applied by passively dorsiflexing the ankle. The angle of dorsiflexion of the ankle at 25 N force shall be recorded and the value obtained noted.
Numeric Pain Rating Scale (1-10 scale) | Change between baseline(immediately before intervention) and post intervention (1 month)
  The numerical pain scale is a unique 11-point numerical scale that has been extensively validated. Pain scores are interpreted as: "0 = no pain"; "1-3 = mild pain"; "4-6 = moderate pain"; "7-10 = severe pain".
Global Rating of Change scale (15 items) | Change between baseline(immediately before intervention) and post intervention (1 month)
  This scale allows us to know the personal evolution experienced by the patient and is considered an efficient way of knowing the score given by the patient to the perceived clinical change. It is a Likert-type scale with 15 items, of which 7 are for improvement, 7 for worsening and 1 for "no change". The patient will be asked to report how he/she felt at the beginning of the treatment; better, worse or no change. If the patient answers better or worse, they will be asked, with the scale in front of them, to indicate whether they are: a little bit almost the same, a little, a little, some, a lot, a lot or very much better or worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain